CLINICAL TRIAL: NCT04486820
Title: Immunohistochemical Study of Chordomas to Improve Their Diagnosis and Prognosis Care
Acronym: CHORDOMES
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Saint Etienne (Other)
Responsible Party: Sponsor
Other Study IDs: 20CH028
Record Dates: First submitted 2020-07-22; First posted 2020-07-27 (Actual); Last update posted 2020-07-27 (Actual); Status verified 2020-07

CONDITIONS: Chordoma
Keywords: Immunohistochemical; PD-L1; CD8; CDX2; INSM1; FOXA1
MeSH Terms: conditions — Chordoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Chordoma: Patients diagnosed with chordoma
  Interventions: Other: Analysis Immunohistochemical

INTERVENTIONS:
Other: Analysis Immunohistochemical — Analysis of histological material for immunohistochemical study. To explore PD-L1, CD8, CDX2, INSM1 and FOXA1 expression

SUMMARY:
Chordomas are very rare malignant tumors, chemo-resistant with high propensity for recurrence. The role of immunotherapy in these patients remains largely unexplored while PD-L1 and CD8 status in the micro-environment of chordomas is basically not known. Similarly, this tumor often poses diagnostic difficulties due to its resemblance with metastasis or chondrosarcoma, thus, it would be useful to know the expression status of factors used during the work-up of metastatic or mesenchymal tumors, like CDX2, INSM1 and FOXA1, which remains unknown for chordomas. Thus, the aim of the study is to explore PD-L1, CD8, CDX2, INSM1 and FOXA1 expression in a series of chordomas and compare it with clinico-pathological and prognostic features.

DETAILED DESCRIPTION:
Retrospective, non-interventional study. A series of chordomas will be analyzed for detailed histologic features and for various immunohistochemical factors and results will be compared with clinical factors, like overall and disease-free survival.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with chordoma
* Sufficient histological material available
* Tumor expression of brachyury

Exclusion Criteria:

- Insufficient histological material

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients diagnosed with chordoma
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2020-04-01 (Actual); Primary Completion 2020-07-01 (Actual); Study Completion 2020-07-01 (Actual)

PRIMARY OUTCOMES:
Expression of PD-L1 | Baseline
  measured by immunohistochemical method
Expression of CD8 | Baseline
  measured by immunohistochemical method
Expression of CDX2 | Baseline
  measured by immunohistochemical method
Expression of INSM1 | Baseline
  measured by immunohistochemical method
Expression of FOXA1 | Baseline
  measured by immunohistochemical method

SECONDARY OUTCOMES:
Histological type of tumor | Baseline
  data collected in personal health records.
Tumor location | Baseline
  data collected in personal health records.
survival of patients after diagnosis with or without progression | Baseline
  data collected in personal health records.

CONTACTS AND LOCATIONS:
Overall Officials: Georgia KARPATHIOU, MD, Principal Investigator — CHU SAINT-ETIENNE
Locations (1):
- CHU de Saint-Etienne, Saint-Etienne, France

IPD SHARING:
Plan to Share IPD: No